CLINICAL TRIAL: NCT00749632
Title: An Open-Label, Dose Escalating Study to Evaluate the Safety of Intravaginal Oxybutynin in Subjects With Urge Urinary Incontinence
Brief Title: A Study of Oxybutynin for the Treatment of Urge Urinary Incontinence
Acronym: FP1097-002
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: FemmePharma Global Healthcare, Inc. (Industry)
Responsible Party: Peter K. Mays, Ph.D. / V.P. Pharmaceutical Development, FemmePharma Global Healthcare, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FP1097-002
Record Dates: First submitted 2008-09-05; First posted 2008-09-09 (Estimated); Last update posted 2009-10-15 (Estimated); Status verified 2009-10

CONDITIONS: Urinary Incontinence, Urge
Keywords: urinary incontinence, urge; urinary urge incontinence; urge incontinence; over active bladder
MeSH Terms: conditions — Urinary Incontinence, Urge | interventions — oxybutynin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator)
  Interventions: Drug: oxybutynin
- 2 (Active Comparator)
  Interventions: Drug: oxybutynin
- 3 (Active Comparator)
  Interventions: Drug: oxybutynin

INTERVENTIONS:
Drug: oxybutynin — low dose oxybutynin administered daily
  Arms: 1
Drug: oxybutynin — middle dose oxybutynin administered daily
  Arms: 2
Drug: oxybutynin — high dose oxybutynin administered daily
  Arms: 3

SUMMARY:
The purpose of this study is to determine the safety of three doses of oxybutynin for the treatment of urge urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Females 18 to 75 years of age
* Has reported symptoms of urge urinary incontinence/overactive bladder

Exclusion Criteria:

* Is pregnant or lactating
* Has had lower urinary tract surgery within 6 months prior to Screening
* Has a history of urinary retention

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2007-07; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Number of micturations and incontinence episodes. | Two weeks pretreatment and three weeks on treatment

CONTACTS AND LOCATIONS:
Overall Officials: Peter K. Mays, Ph.D., Study Director — FemmePharma Global Healthcare, Inc.
Locations (2):
- United States (2):
  - SNBL Clinical Pharmacology Center, Baltimore, Maryland
  - Advanced Biomedical Research, Hackensack, New Jersey